CLINICAL TRIAL: NCT06393348
Title: A Multicenter, Randomized, Double-blinded, Placebo-controlled, Parallel-group Phase ⅡStudy to Evaluate the Efficacy and Safety of HRS-7535 in T2DM Subjects Poorly Controlled With Metformin and SGLT2i.
Brief Title: Efficacy and Safety of HRS-7535 Tablets in T2DM Subjects Poorly Controlled With Metformin and SGLT2i.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HRS-7535-205
Record Dates: First submitted 2024-04-28; First posted 2024-05-01 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Subjects will receive escalated dose of HRS-7535 administered orally
  Interventions: Drug: HRS-7535
- Group B (Experimental): Subjects will receive dose of HRS-7535 administered orally
  Interventions: Drug: HRS-7535
- Group C (Placebo Comparator): Subjects will receive Placebo administered orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HRS-7535 — HRS-7535
  Arms: Group A; Group B
Drug: Placebo — Placebo
  Arms: Group C

SUMMARY:
2 weeks screening period, 3 weeks run-in period, 16 weeks double-blind treatment period, to evaluate the Safety and Efficacy of HRS-7535 in Subjects with Type 2 Diabetes who have Inadequate Glycemic Control on Metformin and SGLT2i.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 18-75 years of age at the time of signing informed consent;
2. Have T2DM (based on the 2020 Chinese Diabetes Society [CDS] diagnostic criteria)
3. HbA1c为7.5%≤HbA1c≤11.0% at the screening visit；
4. FPG≤15 mmol/L at the screening visit;
5. Have been treated with an SGLT2i with metformin, for at least 8 weeks;
6. At screening and random visit, 20.0 ≤BMI≤ 35.0 kg/m2;
7. Able and willing to provide a written informed consent

Exclusion Criteria:

1. Have type 1 diabetesmellitus;
2. History of acute cardiovascular and cerebrovascular diseases within 6 months prior to screening;
3. Any organ-system malignancies developed within 5 years except for cured local basal cell cancer of the skin and in-situ cancer of the cervix;
4. history of blood donation or blood loss in the 3 months before screening, or blood transfusion in the 2 months before screening;
5. Surgery is planned during the trial;
6. Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using an adequate contraceptive method;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2024-05-17 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline at Week 16 | Week 16

SECONDARY OUTCOMES:
Proportion of subjects achieving HbA1c target of <7.0% at 16 weeks | 16 weeks
Proportion of subjects achieving HbA1c target of ≤6.5% at 16 weeks | 16 weeks
The change in fasting blood glucose from baseline to 16 weeks | 16 weeks
The change in in body weight from baseline to 16 weeks | 16 weeks
The change in 7-point SMBG profile from baseline to 16 weeks | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangdong, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided